CLINICAL TRIAL: NCT04725071
Title: Immunonutrition Supplementation for Improved Burn Wound Healing in Older Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1692; A539714 (Other: UW Madison); SMPH/SURGERY/TRAUMA (Other: UW Madison); Protocol Version 1/14/2021 (Other: UW Madison)
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Burn Wound
Keywords: immunonutrition
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunonutrition (Experimental): Participants will consume a 6oz immunonutrition drink 2 times daily for 7 days and then once a day for remaining hospital stay.
  Interventions: Dietary Supplement: Impact Advanced Recovery
- Conventional Supplement (Active Comparator): Participants will consume a 6oz conventional supplement drink 3 times daily for 7 days and then once a day for remaining hospital stay.
  Interventions: Dietary Supplement: Boost High Protein

INTERVENTIONS:
Dietary Supplement: Impact Advanced Recovery — L-arginine and omega-3 rich supplement
  Arms: Immunonutrition
Dietary Supplement: Boost High Protein — conventional supplement
  Arms: Conventional Supplement

SUMMARY:
This pilot study aims to assess the feasibility of providing immunonutrition supplementation to older burn patients (age 55 and older) and its impact on burn wound healing. Supplements containing arginine and omega 3 fatty acids have been shown to have beneficial effects on healing in other types of wounds but data within the burn population remains limited. 20 participants will be randomized into two arms, immunonutrition or conventional supplement and can expect to be on study for 3 months.

DETAILED DESCRIPTION:
Studies performed previously in burn patients have had mixed patient cohorts with small sample sizes and these have failed to show any large improvements in wound healing. However, in older populations the investigators suspect that immunonutrition supplements may have a larger benefit to these patients as they often present with malnutrition and are more likely to struggle with delayed wound healing. In this pilot study, the investigators look to assess the impact of immunonutrition supplements the burn wound healing of adults over the age of 55 years with 1-15% total burn surface area (TBSA) partial thickness and full thickness burn injuries.

The primary outcome objective of the study will be time to complete wound closure. The secondary objectives include need for surgical grafting, length of inpatient stay, and infections including pneumonia, urinary tract infections, wound infections, and blood stream infections.

ELIGIBILITY:
Inclusion Criteria:

* Subject has partial of full thickness thermal injury of 1-15% of total body surface area (TBSA)
* Subject has an inpatient admission for their burn
* Subject or authorized decision maker understands the study procedures and can provide informed consent to participate in the study and authorization for release of relevant protected health information to the study investigator

Exclusion Criteria:

* Subject with inhalation injury and/or intubation
* Subject receiving immunosuppressive medications including chronic steroids, immune modulating medications, and chemotherapy prior to admission
* Subject with pre-existing severe chronic liver disease or end stage renal disease

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Time to Complete Wound Closure | up to 3 months

SECONDARY OUTCOMES:
Incidence of Surgical Grafting | up to 3 months
Length of Inpatient Stay | up to 3 months
Incidence of Infections | up to 3 months
  Infectious complications include pneumonia, urinary tract infection, wound infection, and blood stream infection.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Busch, MD, FACS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT04725071/ICF_000.pdf